CLINICAL TRIAL: NCT02693600
Title: Comparison Between Hemitrapeziectomy and Total Trapeziectomy With Ligament Reconstruction and Tendon Interposition in Trapeziometacarpal Osteoarthritis II-III Eaton-Littler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Ferran Fillat Gomà, MD, MSc, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPTCOT2014/01
Record Dates: First submitted 2016-02-17; First posted 2016-02-26 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Trapeziometacarpal Osteoarthritis
Keywords: Total Trapeziectomy; Partial Trapeziectomy; Ligamentoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Partial Trapeziectomy (PT) (Active Comparator): Patients with Osteoarthritis of the trapeziometacarpal joint determined by the classification of Eaton-Littler (stages II-III) treated with with ligamentoplasty and partial trapeziectomy.
  Interventions: Procedure: Ligamentoplasty with partial trapeziectomy
- Total Trapeziectomy (TT) (Active Comparator): Patients with Osteoarthritis of the trapeziometacarpal joint determined by the classification of Eaton-Littler (stages II-III) treated with ligamentoplasty and total trapeziectomy.
  Interventions: Procedure: Ligamentoplasty with total trapeziectomy

INTERVENTIONS:
Procedure: Ligamentoplasty with partial trapeziectomy
  Arms: Partial Trapeziectomy (PT)
Procedure: Ligamentoplasty with total trapeziectomy
  Arms: Total Trapeziectomy (TT)

SUMMARY:
1. Introduction:

   Investigators think that surgery with preservation of healthy joints (hemitrapeziectomy) in trapeziometacarpal osteoarthritis without affecting sapho-trapezo-trapezoid joints, is better for scaphoid stability by preventing its collapse and thus preserving the stability of the carpus.
2. Objectives and Hypothesis:

   Ligamentoplasty with partial trapeziectomy in grades II-III Eaton presents better results in the pollicis-lateral pinch (key pinch) strength than ligamentoplasty with total trapeziectomy.

   Main Objective:

   To demonstrate using the dynamometer that the postoperative key pinch strength higher using ligamentoplasty with partial trapeziectomy in grades II-III Eaton.

   Secondary objectives:

   To measure the collapse of the first column of thumb using calibrated radiographic analysis. Pain (E.V.A Scale). Range of motion (measured with goniometer). Quality of life (DISABILITIES OF THE ARM, SHOULDER AND HAND questionnaire).
3. Methodology:

It is a single-center randomized trial, parallel-group, in which two types of surgical techniques (TT - TP) will be compared. Patients will be randomized in this two techniques will be followed for one year, in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Osteoarthritis in the trapeziometacarpal joint determined by the classification of Eaton-Littler (stages II-III) with trapeziometacarpal joint pain, loss of function, that were included in surgical waiting list and have accepted under informed consent, including the study.

Exclusion Criteria:

* Patients with osteoarthritis Eaton-Littler (stage IV).
* Patients with huge affection of trapezium subchondral cysts and poor quality of trabecular bone.
* Cognitive impairment.
* Old fracture with impairment of the same extremity.
* Rheumatic active illness.
* Patients who withdraw their informed consent, or in case of impossibility of opinion by clinical status, whose legal guardians or close relatives to withdraw their informed consent to participate in the study.
* Patients who for any reason not related to the indication needed discontinue study participation or impossible to carry out assessments under more than two follow-up visits.
* Patients in whom it is considered that participation in the clinical study can be a prejudice, the physician responsible for patient care opinion.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-09; Primary Completion 2016-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Changes in the pollicis-lateral pinch strength | Before, three Months and One year after surgery.
  In kilograms and measured with dynamometer.

SECONDARY OUTCOMES:
Changes in pain score assessed with E.V.A Scale | Before, three Months and One year after surgery.
  Assessment is performed by E.V.A Scale.
Changes in range of motion | Before, three Months and One year after surgery.
  Opposition, retropulsion and radial abduction were registered.
Changes in Collapse of the first column of thumb using calibrated radiographic analysis | Before, three Months and One year after surgery.
  To measure the collapse of the first column of thumb using calibrated radiographic analysis
Changes in Quality of life assessed with the Disabilities of the arm, shoulder and hand questionnaire (DASH questionnaire) | Before, three Months and One year after surgery.
  Assessment is performed by specific Disabilities of the arm, shoulder and hand questionnaire (DASH questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Ricard Sánchez-Flo, MD, Study Director — Hospital Universitario Parc Taulí de Sabadell; Ferran Fillat-Gomà, MD, Principal Investigator — Hospital Universitario Parc Taulí de Sabadell
Locations (1):
- Hospital Universitario Parc Taulí, Sabadell, Barcelona, Spain